CLINICAL TRIAL: NCT03234049
Title: The Use of a Pediatric Trauma Checklist to Improve Clinical Performance in a Simulated Trauma Resuscitation: a Randomized Trial
Brief Title: The Use of a Pediatric Trauma Checklist to Improve Clinical Performance in a Simulated Trauma Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KidSIM Simulation Program (Network)
Collaborators: KidSIM-ASPIRE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB16-1479
Record Dates: First submitted 2017-01-03; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Trauma
Keywords: pediatric; checklist; cognitive aid
MeSH Terms: conditions — Wounds and Injuries | interventions — Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): In the control arm, teams will not receive a copy of the checklist for use.
- Checklist Arm (Experimental): In the intervention arm, the participants will watch a 10 minute recorded educational video demonstrating the use of the trauma checklist prior to their simulation scenario. These teams will subsequently receive a copy of the checklist for use during their simulation scenario.
  Interventions: Other: Checklist

INTERVENTIONS:
Other: Checklist — The Alberta Children's Hospital Trauma Checklist was developed by the ACH Resuscitation Council Trauma Committee in response to a quality assurance review of high-acuity trauma activations. It is a cognitive aid and focuses in particular on pre-arrival preparation and a pre-departure review prior to patient transfer to diagnostic imaging or the operating room.
  Arms: Checklist Arm

SUMMARY:
The use of a pre-arrival and pre-departure trauma checklist to optimize care has not yet been studied. The Alberta Children's Hospital (ACH) Trauma Checklist was developed by the ACH Resuscitation Council with input from the ACH Trauma Program. The purpose of this study is to determine if the introduction of the ACH Trauma Checklist as a cognitive aid, coupled with an educational session, will improve clinical performance in a simulated environment. The investigators plan to conduct a pilot, randomized control trial assessing the impact of the ACH trauma checklist on time to critical interventions on a simulated pediatric patient by multidisciplinary teams. The investigators hypothesize that teams who use a trauma checklist as a cognitive aid will have faster initiation of key clinical interventions within a simulated pediatric trauma resuscitation. Improvements in performance in a simulated environment with this tool may translate to similar results in the clinical setting.

DETAILED DESCRIPTION:
Research Aims:

Aim 1: To evaluate the effectiveness of a pre-arrival, pre-departure trauma checklist on improving time to initiation of key clinical interventions in a simulated pediatric trauma scenario

Aim 2: To evaluate the impact of a pre-arrival, pre-departure trauma checklist on completion of primary and secondary survey tasks as demonstrated by an Advanced Trauma Life Support (ATLS) performance tool.

Aim 3: To evaluate the cognitive task load of a trauma checklist on emergency department physicians during a simulated trauma resuscitation scenario.

Aim 4: To describe patterns of eye movement of a trauma team leader in a simulated scenario in relation to critical patient interventions and team communication.

METHODS:

POPULATION:

Simulation scenarios will be run with multidisciplinary trauma teams recruited from the Alberta Children's Hospital. Each team will be comprised of a trauma team leader, second physician, three registered nurses and a respiratory therapist. Confederate actors will play the role of the medication nurse and respiratory therapist.

STUDY DESIGN:

This study utilizes a prospective, randomized controlled study design. The investigators propose a randomized control trial methodology with a control group representing standard practice to justify the change to adopt the method amongst clinical trauma teams.

Participants recruited to partake in the study will be asked to perform as members of a pediatric trauma resuscitation team. Each team of healthcare providers will be randomized into one of two study arms. In the intervention arm, the participants will watch a 10-minute recorded educational video demonstrating the use of the trauma checklist prior to their simulation scenario. These teams will subsequently receive a copy of the checklist for use during their simulation scenario. In the control arm, teams will not receive a copy of the checklist for use. All simulated trauma resuscitations will be video recorded and reviewed.

All teams will be asked to participate in a standardized 20-minute trauma resuscitation simulation scenario. This scenario will be followed by a 10-minute debriefing session facilitated by a simulation consultant. Following the trauma resuscitation scenario, and debriefing, the trauma team leader and bedside physician will be asked to complete the NASA Task Load Index (NASA-TLX) survey on cognitive workload. The data collected from this survey, will allow further insight into the impact on mental workload on participants with the use of a cognitive aid.

In addition, the trauma team leader will be asked to wear an eye-tracking device during the simulation scenario. Eye movements are recorded using an eye tracking system. The system captures a scene view calibrated to the participant's perspective of the environment, and an eye view capturing the surface anatomy of the eye (i.e. pupil, iris, sclera, eyelids). The software processes eye and scene data to compute point of gaze data in the environment. Eye-tracking data will be collected and analyzed for development of future studies. In particular, the study investigators aim to describe patterns of eye tracking of a trauma team leader during periods of critical interventions and key team member communication within a simulated scenario.

SAMPLE SIZE & STATISTICAL ANALYSIS:

This study is a pilot study and the investigators will use team performance as unit of measure. In order to achieve a significant level of 0.05 and a power of 0.8, 12 teams per group allows us to detect a large effect size (d = 1.2). A 2-sample t-test is planned to detect the difference in time to initiation of key interventions between 2 groups. If the data does not fall with a normal distribution, the team will use the Wilcoxon rank sum test.

POSSIBLE PROBLEMS & ANTICIPATED SOLUTIONS:

1. Participants may have prior exposure to the trauma checklist: The Alberta Children's Hospital Trauma checklist has been available for use since July 2016. Physical copies are available in the trauma bay; however, the checklist was not formally introduced to the department staff with specific educational initiatives, demonstrations or rounds presentations. Less than 5 completed checklists have been submitted to the Trauma Committee for review. The success of checklist use is influenced by implementation and team culture. The investigators anticipate that participants will have minimal experience with checklist use.
2. Imprecision of outcome measurements: Defining the exact timing of initiation and completion of clinical tasks by video review can be difficult and variable. The research team will determine standardized definitions for video reviewers. All video reviewers will undergo an hour long training session and assessment of their inter-rater reliability.
3. Variability within the simulation scenario: A standardized simulation lab will be prepared. All simulations will be run by a study co-investigator and study coordinator. Confederate actors will undergo specific training and have tightly scripted roles.

Confidentiality and Privacy Protection

Informed and written consent to participate in this research study will be obtained from each team member before the start of each simulation scenario. All data will be stored on a password protected computer within a secured server that can only be accessed by research team members. Data will be destroyed after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Trauma team leader inclusion criteria:

   * Pediatric emergency medicine physician
2. Second physician inclusion criteria:

   * Pediatric emergency medicine physician
3. Nurse inclusion criteria:

   * Pediatric emergency registered nurse

Exclusion criteria:

* Previous participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time measurement interval to initiation of endotracheal tube placement | within the 20 minute simulation scenario
  Interval from start of scenario to endotracheal tube placement
Time measurement interval to initiation of induction medication | within the 20 minute simulation scenario
  Interval from start of scenario to delivery of intubation induction medication
Time measurement interval to initiation of paralytic medication | within the 20 minute simulation scenario
  Interval from start of scenario to delivery of intubation paralytic medication
Time measurement interval to initiation of bag mask ventilation | within the 20 minute simulation scenario
  Interval from start of scenario to first assisted bag mask breath
Time measurement interval to initiation of fluid bolus administration | within the 20 minute simulation scenario
  Interval from start of scenario to initiation of first crystalloid fluid bolus
Time measurement interval to initiation of blood product administration | within the 20 minute simulation scenario
  Interval from start of scenario to initiation of first blood product administration
Time measurement interval to application of pelvic binder | within the 20 minute simulation scenario
  Interval from start of scenario to application of pelvic binder
Time measurement interval to Glasgow Coma Score calculation | within the 20 minute simulation scenario
  Interval from start of scenario to first verbalized and calculated Glasgow Coma Score
Time measurement interval to initiation of hyperosmolar therapy | within the 20 minute simulation scenario
  Interval from start of scenario to initiation of hyperosmolar therapy, either mannitol or 3% saline
Time measurement interval to completion of log roll | within the 20 minute simulation scenario
  Interval from start of scenario to completion of patient log roll

SECONDARY OUTCOMES:
Advanced Trauma Life Support Task Performance | within the 20 minute simulation scenario
  ATLS performance will be scored based on rates of completion of primary and secondary survey tasks, using a previously derived Trauma Resuscitation Checklist
Checklist completion | within the 20 minute simulation scenario
  In the intervention arm, the investigators will determine the completion rate of the ACH trauma checklist by video review.
Eye movements of the trauma team leader | within the 20 minute simulation scenario
  Data will be recorded off an eye tracking device worn by the trauma team leader. In particular, the investigators aim to describe patterns of eye tracking of a trauma team leader during periods critical patient interventions and key team member communication within a simulated scenario. There are 3 specific areas of interest: the patient, the monitor, and the external environment. The frequency of which eye movements rest on those areas will be tracked. This will be reported as a total duration of time (in minutes) spent looking at each of the 3 areas of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, MD FRCPC, Principal Investigator — Alberta Children's Hospital, University of Calgary, KidSIM
Locations (1):
- KidSIM, Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No